CLINICAL TRIAL: NCT01347801
Title: Mechanisms of Insulin Resistance in Critical Illness: Role of Systemic Inflammation and GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kirsten Moller, MD, PH.D, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HS:H-3-2009-108
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Hypoglycaemia
Keywords: GLP-1; Inflammation; Glucose
MeSH Terms: conditions — Hypoglycemia; Inflammation | interventions — Glucagon-Like Peptide 1; Sodium Chloride; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 2C - 1 (Placebo Comparator): TNF and OGTT and saline
  Interventions: Drug: Placebo (Saline); Drug: TNF-alfa; Other: OGTT
- 2C - 2 (Active Comparator): TNF and OGTT and GLP-1
  Interventions: Drug: GLP-1; Drug: TNF-alfa; Other: OGTT
- 2C - 3 (Placebo Comparator): TNF and IVGTT and saline
  Interventions: Drug: Placebo (Saline); Drug: TNF-alfa; Other: IVGTT
- 2C - 4 (Active Comparator): TNF and IVGTT and GLP-1
  Interventions: Drug: GLP-1; Drug: TNF-alfa; Other: IVGTT
- 2A-1 (Placebo Comparator): Saline infusion and OGTT
  Interventions: Drug: Placebo (Saline); Other: OGTT
- 2A-2 (Placebo Comparator): Saline and IVGTT
  Interventions: Drug: Placebo (Saline); Other: IVGTT
- 2A-3 (Active Comparator): TNF and OGTT
  Interventions: Drug: TNF-alfa; Other: OGTT
- 2A-4 (Active Comparator): TNF and IVGTT
  Interventions: Drug: TNF-alfa; Other: IVGTT
- 1C (Experimental): OGTT and corresponding IVGTT
  Interventions: Other: OGTT; Other: IVGTT

INTERVENTIONS:
Drug: GLP-1 — GLP-1 1,2pmol/kg/min i.v. infusion for 4 hours
  Arms: 2C - 2; 2C - 4
Drug: Placebo (Saline) — Normal saline (NaCl 0,9%)
  Arms: 2A-1; 2A-2; 2C - 1; 2C - 3
Drug: TNF-alfa — 1000ng/m2 BSA/hour i.v. infusion for 4-6 hours
  Arms: 2A-3; 2A-4; 2C - 1; 2C - 2; 2C - 3; 2C - 4
Other: OGTT — Oral glucose tolerance test with 75 g glucose
  Arms: 1C; 2A-1; 2A-3; 2C - 1; 2C - 2
Other: IVGTT — Intravenous glucose tolerance test with infusion of 20% glucose matching the glucose profile of the corresponding OGTT
  Arms: 1C; 2A-2; 2A-4; 2C - 3; 2C - 4

SUMMARY:
The purpose of this study is to determine the role of inflammation and the insulin regulating hormone GLP-1 during critical illness.

DETAILED DESCRIPTION:
Critically ill patients often exhibit hyperglycaemia. Although the cause of this hyperglycaemia is probably multifactorial, peripheral insulin resistance is a major contributor, similar to type 2 diabetes mellitus (T2D). There are several similarities between critical illness and T2D, including the presence of systemic inflammation and increased plasma free fatty acids (FFA), all of which may induce insulin resistance in healthy volunteers. In critical illness, elevated catecholamines, cortisol, growth hormone and glucagon may also contribute to insulin resistance.

The degree of hyperglycaemia correlates with mortality in ICU patients. van den Berghe et al. found that IV infusion of insulin to obtain strict normoglycaemia reduced mortality as well as morbidity in critically ill surgical patients and in some medical ICU patients.

However, insulin increases the risk of hypoglycaemia; this is a major obstacle to strict euglycaemia in ICU patients and may explain the inability of others to reproduce the benefits reported by van den Berghe et al. Thus, alternatives to insulin for controlling plasma glucose (PG) in ICU patients are warranted.

Aim:

To study the role of the incretin hormone, glucagon-like peptide (GLP)-1 for glycaemic, metabolic, hormonal and inflammatory profile in

* critically ill patients in the intensive care unit (ICU) and
* healthy volunteers exposed to a standardised systemic inflammation

ELIGIBILITY:
Inclusion Criteria healthy subjects:

* Healthy (assessed by medical history and clinical examination)
* Age 18-40years
* BMI < 30kg/m2

Exclusion Criteria healthy subjects:

* Previous resection of the small intestine (not including the appendix)
* presence of any inflammatory illness during the fortnight preceding the study

Inclusion Criteria critically ill patients:

* Age>18 years
* HbA1C<6,5%
* Admission to the ICU within the last 72 hours

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Substudy 2C (12 Healthy volunteers): GLP-1 | 6 weeks after intervention
  Increased plasma insulin and C-peptide (intact insulinotropic effect of GLP-1) during GLP-1 infusion in healthy volunteers.
Substudy 2A (12 Healthy volunteers): Insulin, C-peptide and incretin hormone response | 6 weeks after intervention
  Insulin, c-peptide and incretin hormone response to glucose stimulation during standardized systemic inflammation (TNF infusion) compared to placebo (saline infusion)
Substudy 1C(8 patients, 8 healthy controls): Insulin, C-peptide and incretin hormone response | 6 weeks after intervention
  Insulin, c-peptide and incretin hormone response to glucose stimulation during IVGTT compared to OGTT in critically ill patients admitted to the ICU

SECONDARY OUTCOMES:
Substudy 2C (12 Healthy volunteers): Clamp | 6 weeks after intervention
  Enhanced insulin response (AUC) and reduced difference between the AUC obtained during OGTT and IGGTT (reduced endogenous incretin effect) during an isoglycaemic intravenous glucose tolerance test (IVGTT) in healthy volunteers receiving TNF-infusion.
Substudy 2A (12 Healthy volunteers): The incretin effect | 6 weeks after intervention
  The difference between the plasma insulin AUC obtained during OGTT and IVGTT (endogenous incretin effect).
Substudy 1C (8 patients, 8 healthy controls): The incretin effect | 6 weeks after intervention
  The difference between the plasma insulin AUC obtained during OGTT and IVGTT (endogenous incretin effect)in non-diabetic critically ill patients admitted to the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Møller, MD, Ph.D., DMSc, Principal Investigator — Centre of Inflammation and Metabolism
Locations (2):
- Denmark (2):
  - Centre of Inflammation and Metabolism - Rigshospitalet 7641, Copenhagen
  - University of Copenhagen, Copenhagen

REFERENCES:
- [Background] McCowen KC, Malhotra A, Bistrian BR. Stress-induced hyperglycemia. Crit Care Clin. 2001 Jan;17(1):107-24. doi: 10.1016/s0749-0704(05)70154-8. PMID 11219223
- [Background] Mizock BA. Alterations in fuel metabolism in critical illness: hyperglycaemia. Best Pract Res Clin Endocrinol Metab. 2001 Dec;15(4):533-51. doi: 10.1053/beem.2001.0168. PMID 11800522
- [Background] Rusavy Z, Sramek V, Lacigova S, Novak I, Tesinsky P, Macdonald IA. Influence of insulin on glucose metabolism and energy expenditure in septic patients. Crit Care. 2004 Aug;8(4):R213-20. doi: 10.1186/cc2868. Epub 2004 May 26. PMID 15312220
- [Background] Beal AL, Cerra FB. Multiple organ failure syndrome in the 1990s. Systemic inflammatory response and organ dysfunction. JAMA. 1994 Jan 19;271(3):226-33. PMID 8080494
- [Background] Schmidt MI, Duncan BB, Sharrett AR, Lindberg G, Savage PJ, Offenbacher S, Azambuja MI, Tracy RP, Heiss G. Markers of inflammation and prediction of diabetes mellitus in adults (Atherosclerosis Risk in Communities study): a cohort study. Lancet. 1999 May 15;353(9165):1649-52. doi: 10.1016/s0140-6736(99)01046-6. PMID 10335783
- [Background] Wolfe RR, Martini WZ. Changes in intermediary metabolism in severe surgical illness. World J Surg. 2000 Jun;24(6):639-47. doi: 10.1007/s002689910105. PMID 10773115
- [Background] Boden G, Shulman GI. Free fatty acids in obesity and type 2 diabetes: defining their role in the development of insulin resistance and beta-cell dysfunction. Eur J Clin Invest. 2002 Jun;32 Suppl 3:14-23. doi: 10.1046/j.1365-2362.32.s3.3.x. PMID 12028371
- [Background] Thijs LG, Hack CE. Time course of cytokine levels in sepsis. Intensive Care Med. 1995 Nov;21 Suppl 2:S258-63. doi: 10.1007/BF01740764. PMID 8636533
- [Background] Krogh-Madsen R, Plomgaard P, Moller K, Mittendorfer B, Pedersen BK. Influence of TNF-alpha and IL-6 infusions on insulin sensitivity and expression of IL-18 in humans. Am J Physiol Endocrinol Metab. 2006 Jul;291(1):E108-14. doi: 10.1152/ajpendo.00471.2005. Epub 2006 Feb 7. PMID 16464907
- [Background] Roden M, Price TB, Perseghin G, Petersen KF, Rothman DL, Cline GW, Shulman GI. Mechanism of free fatty acid-induced insulin resistance in humans. J Clin Invest. 1996 Jun 15;97(12):2859-65. doi: 10.1172/JCI118742. PMID 8675698
- [Background] Voerman BJ, Strack van Schijndel RJ, Groeneveld AB, de Boer H, Nauta JP, Thijs LG. Effects of human growth hormone in critically ill nonseptic patients: results from a prospective, randomized, placebo-controlled trial. Crit Care Med. 1995 Apr;23(4):665-73. doi: 10.1097/00003246-199504000-00014. PMID 7712756
- [Background] Finney SJ, Zekveld C, Elia A, Evans TW. Glucose control and mortality in critically ill patients. JAMA. 2003 Oct 15;290(15):2041-7. doi: 10.1001/jama.290.15.2041. PMID 14559958
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Van den Berghe G, Wilmer A, Hermans G, Meersseman W, Wouters PJ, Milants I, Van Wijngaerden E, Bobbaers H, Bouillon R. Intensive insulin therapy in the medical ICU. N Engl J Med. 2006 Feb 2;354(5):449-61. doi: 10.1056/NEJMoa052521. PMID 16452557
- [Background] Brunkhorst FM, Engel C, Bloos F, Meier-Hellmann A, Ragaller M, Weiler N, Moerer O, Gruendling M, Oppert M, Grond S, Olthoff D, Jaschinski U, John S, Rossaint R, Welte T, Schaefer M, Kern P, Kuhnt E, Kiehntopf M, Hartog C, Natanson C, Loeffler M, Reinhart K; German Competence Network Sepsis (SepNet). Intensive insulin therapy and pentastarch resuscitation in severe sepsis. N Engl J Med. 2008 Jan 10;358(2):125-39. doi: 10.1056/NEJMoa070716. PMID 18184958
- [Background] Cryer PE. Hypoglycaemia: the limiting factor in the glycaemic management of the critically ill? Diabetologia. 2006 Aug;49(8):1722-5. doi: 10.1007/s00125-006-0306-4. No abstract available. PMID 16758178
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] Holst JJ, Gromada J. Role of incretin hormones in the regulation of insulin secretion in diabetic and nondiabetic humans. Am J Physiol Endocrinol Metab. 2004 Aug;287(2):E199-206. doi: 10.1152/ajpendo.00545.2003. PMID 15271645
- [Background] Kolligs F, Fehmann HC, Goke R, Goke B. Reduction of the incretin effect in rats by the glucagon-like peptide 1 receptor antagonist exendin (9-39) amide. Diabetes. 1995 Jan;44(1):16-9. doi: 10.2337/diab.44.1.16. PMID 7813808
- [Background] Holst JJ. The physiology of glucagon-like peptide 1. Physiol Rev. 2007 Oct;87(4):1409-39. doi: 10.1152/physrev.00034.2006. PMID 17928588
- [Background] Orskov C, Holst JJ, Nielsen OV. Effect of truncated glucagon-like peptide-1 [proglucagon-(78-107) amide] on endocrine secretion from pig pancreas, antrum, and nonantral stomach. Endocrinology. 1988 Oct;123(4):2009-13. doi: 10.1210/endo-123-4-2009. PMID 2901341
- [Background] Creutzfeldt WO, Kleine N, Willms B, Orskov C, Holst JJ, Nauck MA. Glucagonostatic actions and reduction of fasting hyperglycemia by exogenous glucagon-like peptide I(7-36) amide in type I diabetic patients. Diabetes Care. 1996 Jun;19(6):580-6. doi: 10.2337/diacare.19.6.580. PMID 8725855
- [Background] Willms B, Idowu K, Holst JJ, Creutzfeldt W, Nauck MA. Overnight GLP-1 normalizes fasting but not daytime plasma glucose levels in NIDDM patients. Exp Clin Endocrinol Diabetes. 1998;106(2):103-7. doi: 10.1055/s-0029-1211959. PMID 9628239
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Vilsboll T, Krarup T, Deacon CF, Madsbad S, Holst JJ. Reduced postprandial concentrations of intact biologically active glucagon-like peptide 1 in type 2 diabetic patients. Diabetes. 2001 Mar;50(3):609-13. doi: 10.2337/diabetes.50.3.609. PMID 11246881
- [Background] Vilsboll T, Toft-Nielsen MB, Krarup T, Madsbad S, Dinesen B, Holst JJ. Evaluation of beta-cell secretory capacity using glucagon-like peptide 1. Diabetes Care. 2000 Jun;23(6):807-12. doi: 10.2337/diacare.23.6.807. PMID 10841001
- [Background] Knop FK, Vilsboll T, Larsen S, Madsbad S, Holst JJ, Krarup T. No hypoglycemia after subcutaneous administration of glucagon-like peptide-1 in lean type 2 diabetic patients and in patients with diabetes secondary to chronic pancreatitis. Diabetes Care. 2003 Sep;26(9):2581-7. doi: 10.2337/diacare.26.9.2581. PMID 12941722
- [Background] Meier JJ, Weyhe D, Michaely M, Senkal M, Zumtobel V, Nauck MA, Holst JJ, Schmidt WE, Gallwitz B. Intravenous glucagon-like peptide 1 normalizes blood glucose after major surgery in patients with type 2 diabetes. Crit Care Med. 2004 Mar;32(3):848-51. doi: 10.1097/01.ccm.0000114811.60629.b5. PMID 15090972
- [Background] Sokos GG, Bolukoglu H, German J, Hentosz T, Magovern GJ Jr, Maher TD, Dean DA, Bailey SH, Marrone G, Benckart DH, Elahi D, Shannon RP. Effect of glucagon-like peptide-1 (GLP-1) on glycemic control and left ventricular function in patients undergoing coronary artery bypass grafting. Am J Cardiol. 2007 Sep 1;100(5):824-9. doi: 10.1016/j.amjcard.2007.05.022. Epub 2007 Jun 14. PMID 17719327
- [Background] Deane AM, Summers MJ, Zaknic AV, Chapman MJ, Fraser RJ, Di Bartolomeo AE, Wishart JM, Horowitz M. Exogenous glucagon-like peptide-1 attenuates the glycaemic response to postpyloric nutrient infusion in critically ill patients with type-2 diabetes. Crit Care. 2011;15(1):R35. doi: 10.1186/cc9983. Epub 2011 Jan 21. PMID 21255422
- [Background] Deane AM, Chapman MJ, Fraser RJ, Summers MJ, Zaknic AV, Storey JP, Jones KL, Rayner CK, Horowitz M. Effects of exogenous glucagon-like peptide-1 on gastric emptying and glucose absorption in the critically ill: relationship to glycemia. Crit Care Med. 2010 May;38(5):1261-9. doi: 10.1097/CCM.0b013e3181d9d87a. PMID 20228679
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Rosenvinge A, Krogh-Madsen R, Baslund B, Pedersen BK. Insulin resistance in patients with rheumatoid arthritis: effect of anti-TNFalpha therapy. Scand J Rheumatol. 2007 Mar-Apr;36(2):91-6. doi: 10.1080/03009740601179605. PMID 17476613
- [Derived] Nielsen ST, Janum S, Krogh-Madsen R, Solomon TP, Moller K. The incretin effect in critically ill patients: a case-control study. Crit Care. 2015 Nov 16;19:402. doi: 10.1186/s13054-015-1118-z. PMID 26567860
- [Derived] Lehrskov-Schmidt L, Lehrskov-Schmidt L, Nielsen ST, Holst JJ, Moller K, Solomon TP. The effects of TNF-alpha on GLP-1-stimulated plasma glucose kinetics. J Clin Endocrinol Metab. 2015 Apr;100(4):E616-22. doi: 10.1210/jc.2014-4244. Epub 2015 Feb 12. PMID 25675385